CLINICAL TRIAL: NCT02291510
Title: A Randomized, Crossover Study Assessing the Pharmacokinetics of EFB0027 Versus ETB0015 and ETB0014 in Healthy Subjects
Brief Title: Assessing the PK of Met DR, Met IR, and Met XR in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elcelyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LCRM103
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Results first posted 2015-09-21 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 500 mg Met DR BID (Experimental): Two doses of 500 mg metformin delayed-release
  Interventions: Drug: Met DR
- 1000 mg Met DR BID (Experimental): Two doses of 1000 mg metformin delayed-release
  Interventions: Drug: Met DR
- 1000 mg Met IR BID (Active Comparator): Two doses of 1000 mg metformin immediate-release
  Interventions: Drug: Met IR
- 2000 mg Met XR QD (Active Comparator): Single dose of 2000 mg metformin extended-release
  Interventions: Drug: Met XR

INTERVENTIONS:
Drug: Met DR — metformin delayed-release tablets
  Arms: 1000 mg Met DR BID; 500 mg Met DR BID
Drug: Met XR — metformin extended-release tablets
  Arms: 2000 mg Met XR QD
Drug: Met IR — metformin immediate-release tablets
  Arms: 1000 mg Met IR BID

SUMMARY:
This study compared the pharmacokinetics (PK) and assessed the safety of delayed-release metformin (Met DR, EFB0027) at two dosage levels, immediate-release metformin (Met IR, ETB0015), and extended-release metformin (Met XR, ETB0014) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 19 to 65 (inclusive) years old at Visit 1 (Screening)
2. Male, or if female and met all of the following criteria:

   1. Not breastfeeding
   2. Negative pregnancy test result at Visit 1 (Screening) (not applicable to hysterectomized females)
   3. Surgically sterile, postmenopausal, or if of childbearing potential, practiced and was willing to continue to practice appropriate birth control during the entire duration of the study
3. Body mass index (BMI) of 25.0 to 35.0 kg/m² (inclusive) at Visit 1 (Screening)
4. Had a physical examination with no clinically significant abnormalities as judged by the investigator
5. Had normal renal function with an estimated glomerular filtration rate (eGFR) ≥90 mL/min/1.73 m² based on the Modification of Diet in Renal Disease (MDRD) equation
6. Ability to understand and willingness to adhere to protocol requirements

Exclusion Criteria:

1. Had a clinically significant medical condition as judged by the investigator that could potentially affect study participation and/or personal well-being, including but not limited to the following conditions:

   1. Hepatic disease
   2. Gastrointestinal disease
   3. Endocrine disorder (including diabetes and impaired glucose tolerance)
   4. Cardiovascular disease
   5. Central nervous system diseases
   6. Psychiatric or neurological disorders
   7. Organ transplantation
   8. Chronic or acute infection
   9. Orthostatic hypotension, fainting spells or blackouts
   10. Allergy or hypersensitivity
2. Had any chronic disease requiring medication that was adjusted in the past 90 days (subjects could take acute intermittent over-the-counter medications such as Tylenol, if needed)
3. Had major surgery of any kind within 6 months of Visit 1 (Screening)
4. Had a history of >6 kg weight change within 3 months of Visit 1 (Screening)
5. Had clinical laboratory test (clinical chemistry, hematology, or urinalysis) abnormalities judged by the investigator to be clinically significant at Visit 1 (Screening)
6. Had a physical, psychological, or historical finding that, in the investigator's opinion, would make the subject unsuitable for the study
7. Had any drug treatment that affects gastric pH (prescription or over-the-counter), including any antacids or medications such as Rolaids or Pepcid within 2 days of Visit 1 (Screening)
8. Currently abused drugs or alcohol or had a history of abuse that in the investigator's opinion would cause the individual to be noncompliant with study procedures
9. Smoked more than 10 cigarettes per day, 3 cigars per day, 3 pipes per day, used more than 1 can of smokeless tobacco per week, or used a combination of tobacco products that approximate nicotine doses equivalent to 10 cigarettes per day
10. Had donated blood within 3 months of the date of the first dose of randomized study medication, or was planning to donate blood during the study
11. Had received any investigational drug within 2 months (or five half-lives of the investigational drug, whichever was greater) of the date of the first dose of randomized study medication
12. Had known allergies or hypersensitivity to any component of study treatment
13. Was employed by Elcelyx Therapeutics, Inc (that is an employee, temporary contract worker, or designee of the company)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rasmussen, MD, Principal Investigator — Celerion

REFERENCES:
- [Background] DeFronzo RA, Buse JB, Kim T, Skare S, Baron A, Fineman M, editors. Dissociation between Metformin Plasma Exposure and its Glucose-Lowering Effect: A Novel Gut-Mediated Mechanism of Action. 73rd Annual Scientific Meeting of The American Diabetes Association; 2013 June 21-25th; Chicago, Il.
- [Background] Buse JB, DeFronzo RA, Rosenstock J, Kim T, Burns C, Skare S, Baron A, Fineman M. The Primary Glucose-Lowering Effect of Metformin Resides in the Gut, Not the Circulation: Results From Short-term Pharmacokinetic and 12-Week Dose-Ranging Studies. Diabetes Care. 2016 Feb;39(2):198-205. doi: 10.2337/dc15-0488. Epub 2015 Aug 18. PMID 26285584

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: ABDC; Sequence 2: BCAD; Sequence 3: CDBA; Sequence 4: DACB: Treatment A = 1000 mg Met IR BID Treatment B = 500 mg Met DR BID Treatment C = 1000 mg Met DR BID Treatment D = 2000 mg Met XR QD
Period: Overall Study
Arm/Group | Sequence 1: ABDC | Sequence 2: BCAD | Sequence 3: CDBA | Sequence 4: DACB
Started | 5 | 5 | 5 | 5
Completed Treatment A | 5 | 5 | 5 | 5
Completed Treatment B | 5 | 5 | 5 | 4
Completed Treatment C | 5 | 5 | 5 | 4
Completed Treatment D | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 4
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized (ITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: ABDC | Sequence 2: BCAD | Sequence 3: CDBA | Sequence 4: DACB | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (13.6) | 34.8 (13.1) | 33.8 (9.2) | 25.8 (5.0) | 32.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 4 | 6
  Male | 4 | 5 | 4 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 4 | 5 | 5 | 3 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2 | 4
  White | 4 | 3 | 4 | 2 | 13
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.1 (4.0) | 29.5 (2.8) | 28.7 (2.8) | 30.0 (1.8) | 29.6 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: AUC (0-t) of Plasma Metformin
Description: AUC (0-t) = Area under the curve from the time of dosing (0 h) to the time of the last quantifiable concentration after the standardized dinner. Doses were administered 1 min prior to 0 h (standardized dinner) for once daily in the evening (qPM) and twice daily (BID) dosing and 1 min prior to 12 h (standardized breakfast) for once daily in the morning (qAM) and BID dosing.
Time Frame: Time points to create AUC (0-t) were: t = -0.08, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 11, 11.92, 12.5, 13, 13.5, 14, 14.5, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours relative to the start time of the standardized dinner.
Population: Evaluable Population
Measure: Mean (Standard Error); unit: ng*h/mL
Arm/Group | 500 mg Met DR BID | 1000 mg Met DR BID | 1000 mg Met IR BID | 2000 mg Met XR QD
Number analyzed (Participants) | 19 | 19 | 19 | 19
ng*h/mL | 6164 (465) | 9014 (610) | 18709 (1044) | 16989 (968)
Statistical Analysis 1: Comparison: 500 mg Met DR BID vs 2000 mg Met XR QD; 2000 mg Met XR QD is the denominator for the % ratio of least squares (LS) means and the comparator for the p-values; Test type: Superiority or Other; p < 0.001, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 35.4, 90% CI 2-sided [32.27 to 38.74]
Statistical Analysis 2: Comparison: 1000 mg Met DR BID vs 2000 mg Met XR QD; 2000 mg Met XR QD is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p < 0.001, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 52.3, 90% CI 2-sided [47.77 to 57.36]
Statistical Analysis 3: Comparison: 500 mg Met DR BID vs 1000 mg Met IR BID; 1000 mg Met IR BID is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p < 0.001, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 32.1, 90% CI 2-sided [29.30 to 35.18]
Statistical Analysis 4: Comparison: 1000 mg Met DR BID vs 1000 mg Met IR BID; 1000 mg Met IR BID is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p < 0.001, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 47.5, 90% CI 2-sided [43.38 to 52.09]
Statistical Analysis 5: Comparison: 1000 mg Met IR BID vs 2000 mg Met XR QD; 2000 mg Met XR QD is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0832, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 110.1, 90% CI 2-sided [100.50 to 120.68]

2. Primary Outcome: Cmax of Plasma Metformin
Description: Cmax = Maximum concentration from the first dose of study medication administration (0 h) to the time of the last quantifiable concentration following dose administration. Doses were administered 1 min prior to 0 h (standardized dinner) for qPM and BID dosing and 1 min prior to 12 h (standardized breakfast) for qAM and BID dosing.
Time Frame: Time points to create Cmax were: t = -0.08, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 9, 10, 11, 11.92, 12.5, 13, 13.5, 14, 14.5, 15, 16, 17, 18, 19, 20, 21, 22, 23, and 24 hours relative to the start time of the standardized dinner.
Population: Evaluable Population
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | 500 mg Met DR BID | 1000 mg Met DR BID | 1000 mg Met IR BID | 2000 mg Met XR QD
Number analyzed (Participants) | 19 | 19 | 19 | 19
ng/mL | 607 (33) | 905 (56) | 1328 (63) | 1688 (97)
Statistical Analysis 1: Comparison: 500 mg Met DR BID vs 2000 mg Met XR QD; 2000 mg Met XR QD is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p < 0.001, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 35.9, 90% CI 2-sided [32.43 to 39.77]
Statistical Analysis 2: Comparison: 1000 mg Met DR BID vs 2000 mg Met XR QD; 2000 mg Met XR QD is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p < 0.001, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 53.0, 90% CI 2-sided [47.88 to 58.71]
Statistical Analysis 3: Comparison: 500 mg Met DR BID vs 1000 mg Met IR BID; 1000 mg Met IR BID is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p < 0.001, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 45.3, 90% CI 2-sided [40.88 to 50.13]
Statistical Analysis 4: Comparison: 1000 mg Met DR BID vs 1000 mg Met IR BID; 1000 mg Met IR BID is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p < 0.001, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 66.8, 90% CI 2-sided [60.34 to 74.00]
Statistical Analysis 5: Comparison: 1000 mg Met IR BID vs 2000 mg Met XR QD; 2000 mg Met XR QD is the denominator for the % ratio of LS means and the comparator for the p-values; Test type: Superiority or Other; p = 0.0004, ANOVA; Included treatment, sequence, and period and as fixed effects and subject nested within sequence as a random effect; % Ratio of LS Means = 79.3, 90% CI 2-sided [71.65 to 87.86]

ADVERSE EVENTS:
Time Frame: Approximately 18 to 57 days depending on the number of days between the start of Visit 1 and Visit 2 and the number of washout days between the treatment visits
Arm/Group | 500 mg Met DR BID | 1000 mg Met DR BID | 1000 mg Met IR BID | 2000 mg Met XR QD
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/19 | 3/19 | 5/20 | 10/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 500 mg Met DR BID (N=19) | 1000 mg Met DR BID (N=19) | 1000 mg Met IR BID (N=20) | 2000 mg Met XR QD (N=20)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Catheter Site Pain (General disorders) | 1 | 0 | 1 | 1
Catheter Site Related Reaction (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1
Vessel Puncture Site Haematoma (General disorders) | 0 | 0 | 0 | 1
Vessel Puncture Site Pain (General disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study may be published by INSTITUTE, however the publication shall not disclose any SPONSOR Confidential Information, the INSTITUTE shall send the SPONSOR a copy of any such proposed publication 90 days prior to submission for publication, the INSTITUTE, on request of the SPONSOR, shall delete any SPONSOR Confidential Information in the proposed publication, and the INSTITUTE shall, on the SPONSOR's request, delay submission while the SPONSOR files applications for patents.